CLINICAL TRIAL: NCT03563898
Title: Feasibility and Safety in the Management of Fluid Overload in Peritoneal Dialysis Patients Through Sweat Stimulation With the Use of Portable Sauna Bath, Pilot Study
Acronym: SWEAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Pablo Maggiani Aguilera, Principal Investigator, Hospital Civil de Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2222
Record Dates: First submitted 2018-05-23; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-05

CONDITIONS: Fluid Overload; Peritoneal Dialysis Complication
MeSH Terms: conditions — Edema | interventions — Sweating

STUDY DESIGN:
Intervention Model Description: Patients will be subjected daily for 30 minutes to the Portable Sauna Care steam bath (45 degree C temperature). The patient will decide if the time and / or temperature of the Sauna Bath is reduced to Tolerance. Before being subjected to the sauna bath, blood pressure will be taken 10 minutes prior. Weigh the patient with a Scale. You will be informed of the symptoms that may occur during the bath, and if present, you will let the health staff know that you will be present at all times during the bathing period, which will have a SURVEILLANCE TABLE which It will be filled during the intervention where they are monitored and comply with the stipulated norms as well as notes for adverse effects. After the completion of the bath, there will be a space of 15 minutes for the patient to dry the skin and the bathing suit with a towel. After 15 minutes, the patient will be weighed and the blood pressure will be taken again.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sweating with Portable Sauna Bath — Patients will be subjected daily for 30 minutes to the Portable Sauna Care steam bath (45 degree C temperature). The patient will decide if the time and / or temperature of the Sauna Bath is reduced to Tolerance. Before being subjected to the sauna bath, blood pressure will be taken 10 minutes prior. Weigh the patient with a Scale. You will be informed of the symptoms that may occur during the bath, and if present, you will let the health staff know that you will be present at all times during the bathing period, which will have a SURVEILLANCE TABLE which It will be filled during the intervention where they are monitored and comply with the stipulated norms as well as notes for adverse effects. After the completion of the bath, there will be a space of 15 minutes for the patient to dry the skin and the bathing suit with a towel. After 15 minutes, the patient will be weighed and the blood pressure will be taken again.

SUMMARY:
The objective of this pilot study is to evaluate the feasibility and safety of the use of diaphoresis achieved through the use of portable sauna baths in peritoneal dialysis patients with fluid overload

DETAILED DESCRIPTION:
Fluid overload is a common problem in peritoneal dialysis (PD) patients and it is associated with left ventricular hypertrophy and other adverse cardiac consequences. Fluid management is therefore an important aspect in the management of dialysis patient. Despite improvements in dialysis methods and other techniques in these patients, fluid overload persists due to the great limitations of the affected population: physiopathological, economic, educational, social and psychological. The above creates the need for other therapies that lead to the reduction of overload and thus avoid the comorbidity that this entails. The objective of this study is to evaluate the feasibility and safety of the use of diaphoresis achieved through the use of portable sauna baths in peritoneal dialysis patients with fluid overload. The patients are subjected to a period of data collection for 3 days and then use the portable sauna bath 30 minutes a day supervised by the research team during the 6 following days, without interrupting their peritoneal dialysis therapy. We plan to recruit at least 9 patients with PD with fluid overload. Changes in the degree of overhydration are determined by bioimpedance spectroscopy and patient weight at the beginning and end after treatment. Changes in body weight, blood pressure, potassium, urea and creatinine levels, the degree of edema, as well as knowledge about the salt and liquid line were also evaluated. Adverse events will be reported.

ELIGIBILITY:
Inclusion Criteria:

Being on chronic peritoneal dialysis every day since at least 3 months Diagnostic of Fluid overload Stable clinical condition Written informed consent

Exclusion Criteria:

Any cardiovascular event in the last 12 months (acute myocardial infarction, NYHA Heart Failure III-IV, Cardiac Arrhythmia, Cerebral Vascular Event, Unstable-Stable Angina) Peritonitis Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events (grade 2 or above) as measured by CTCAE v 4.0 | Through Day 10 of follow up
  Discontinuation criteria for CTCAE v 4.0 were grade ≥3 adverse events and even grade ≤2 adverse events if the participant wished to withdraw from the study

SECONDARY OUTCOMES:
Degree of overhydration | Through Day 10 of follow up
  The difference at the beginning and the end of overhydration (OH) measured by Bioimpedance, during the duration of the study
Decrease in patient's weight | Through Day 10 of follow up
  The difference of median weight (kg) between control and intervention fase during the duration of the study
Decrease in blood pressure | Through Day 10 of follow up
  The difference of median systolic/diastolic pressure (mmHg) between control and intervention fase during the duration of the study
Decrease in the control of Urea, Creatinine, phosphorus, potassium and calcium levels | Through Day 10 of follow up
  The difference at the beginning and the end of Urea, Creatinine, phosphorus, potassium and calcium serum levels during the duration of the study
Decrease in fluid overload symptoms | Through Day 10 of follow up
  The difference at the beginning and the end of The New York Heart Association (NYHA) Functional Classification of breathlessness (during the duration of the study
Changes in sleep quality | Through Day 10 of follow up
  The difference at the beginning and the end of the Sleep Quality Assessment (PSQI) during the duration of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hosptal Civil Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Derived] Maggiani-Aguilera P, Chavez-Iniguez JS, Navarro-Blackaller G, Hernandez-Morales K, Geraldo-Ozuna AL, Alcantar-Villin L, Montoya-Montoya O, Luquin-Arellano VH, Garcia-Garcia G. Portable sauna stimulated-diaphoresis for the treatment of fluid-overload in peritoneal dialysis patients: A pilot study. Front Med (Lausanne). 2022 Sep 20;9:887609. doi: 10.3389/fmed.2022.887609. eCollection 2022. PMID 36203760